CLINICAL TRIAL: NCT03955705
Title: Analgesic Effectiveness of Nefopam in Patients Undergoing Anterior Cervical Spine Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Si204/2019
Record Dates: First submitted 2019-05-07; First posted 2019-05-20 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Cervical Spine Degeneration
MeSH Terms: interventions — Nefopam; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nefopam (Experimental): Nefopam: 20 mg (infuse at least 15 minutes) every 4-6 hours, max 120 mg/day
  Interventions: Drug: Nefopam 20 mg/ml
- Normal saline solution (Placebo Comparator): Normal saline or 0.9% Sodium Chloride (NaCl) or NSS
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Nefopam 20 mg/ml — Nefopam is a benzoxazocine derivative which is non-opioid and non NSAIDs. The previous studies showed that nefopam can inhibit reuptake of serotonin, norepinephrine and dopamine.
  Other Names: Acupan
  Arms: Nefopam
Drug: Normal saline — 0.9% Sodium chloride (normal saline or NSS)
  Other Names: 0.9% NaCl or NSS
  Arms: Normal saline solution

SUMMARY:
Nefopam is a benzoxazocine derivative which is non-opioid and non NSAIDs. The previous studies showed that nefopam can inhibit reuptake of serotonin, norepinephrine and dopamine. It has no respiratory depression so may be useful in potential airway compromized surgery like anterior cervical discectomy and fusion (ACDF). This study aims to study the analgesic properties of nefopam after ACDF.

DETAILED DESCRIPTION:
The investigators enroll 50 patient who admitted for ACDF. Standard general anesthesia will be performed in all of the patients. Then, an hour before finishing operation, the patients will be divided into two groups. The first group will receive Nefopam 20 mg infuse for 60 min. The another group or group NSS will receive the same amount of 0.9% sodium chloride. The recorded data include patient demographic data, intraoperative blood loss, hemodynamics and pre and postoperative pain scores and Thai version of the Neuropathic Pain Symptom Inventory (NPSI-T score).

ELIGIBILITY:
Inclusion Criteria:

* Patients with cervical spondylosis or cervical spondylotic myelopathy undergoing elective anterior cervical spine surgery such as ACDF or anterior cervical corpectomy and fusion (ACCF)
* American Society of Anesthesiologists (ASA) class I-III
* Age 18-75 years old
* Body weight > 50 kg, BMI < 30 kg/m2

Exclusion Criteria:

* Convulsion or seizure
* Myocardial ischemia or infarction
* Risk of urinary retention from urethral disease or prostate disease
* Angle closure glaucoma
* Patients on monoamine oxidase inhibitor
* Psychiatric patients
* Pregnant or lactated woman
* Creatinine clearance < 30 ml/min
* Allergic to nefopam
* Patients on pregabaline or gabapentin
* Poorly controlled hypertension
* Cannot understand or do the questionnaire of Thai version of Neuropathic pain symptom inventory (NPSI-T) score

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Total morphine consumption | 24 hours
  Intravenous morphine was given to all by patient controlled analgesia (PCA) machine. The higher morphine consumption reflects higher postoperative pain.

SECONDARY OUTCOMES:
The change in Thai version of the Neuropathic Pain Symptom Inventory (NPSI-T score) | 30 days
  Changes in NPSI-T (minimum 0- maximum 100) period by recording NPSI-T at preoperative period, compared with postoperative day 1, 3, 15,30. The total score is 100, the higher scores reflect higher neuropathic pain
The change in pain scores | 72 hours
  Changes in pain scores (minimum 0- maximum 10) at different time point 0 (upon arrival to recovery room), postoperative at 4, 8, 12, 16, 24, 48, 72 hours. The higher scores reflect higher pain.

CONTACTS AND LOCATIONS:
Overall Officials: Manee Raksakietisak, MD, Principal Investigator — Mahidol University
Locations (1):
- Siriraj Hospital Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rao R. Neck pain, cervical radiculopathy, and cervical myelopathy: pathophysiology, natural history, and clinical evaluation. J Bone Joint Surg Am. 2002 Oct;84(10):1872-81. doi: 10.2106/00004623-200210000-00021. No abstract available. PMID 12377921
- [Background] Dordoni PL, Della Ventura M, Stefanelli A, Iannace E, Paparella P, Rocca B, Accorra F. Effect of ketorolac, ketoprofen and nefopam on platelet function. Anaesthesia. 1994 Dec;49(12):1046-9. doi: 10.1111/j.1365-2044.1994.tb04352.x. PMID 7864317
- [Background] Sunshine A, Laska E. Nefopam and morphine in man. Clin Pharmacol Ther. 1975 Nov;18(5 Pt 1):530-4. doi: 10.1002/cpt1975185part1530. PMID 1102231
- [Result] Kim KH, Abdi S. Rediscovery of nefopam for the treatment of neuropathic pain. Korean J Pain. 2014 Apr;27(2):103-11. doi: 10.3344/kjp.2014.27.2.103. Epub 2014 Mar 28. PMID 24748937
- [Result] Martinez V, Beloeil H, Marret E, Fletcher D, Ravaud P, Trinquart L. Non-opioid analgesics in adults after major surgery: systematic review with network meta-analysis of randomized trials. Br J Anaesth. 2017 Jan;118(1):22-31. doi: 10.1093/bja/aew391. PMID 28039239